CLINICAL TRIAL: NCT00101465
Title: Partnership Programs to Reduce Cardiovascular Disparities - Heart Failure Disparities in Native Hawaiians
Brief Title: Partnership Programs for Reducing Cardiovascular Disparities in Native Hawaiians
Status: Completed | Type: Observational
Sponsor: University of Hawaii (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Nobumi Nakamura, University of Hawaii at Manoa
Other Study IDs: 1281; U01HL079163 (NIH)
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
Keywords: Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to improve cardiovascular disease (CVD) outcomes in racial and ethnic minorities in Hawaii.

DETAILED DESCRIPTION:
BACKGROUND:

While there has been great progress in reducing CVD morbidity and mortality in the U.S. over the past 40 years, some minority groups have not benefitted from this progress, and continue to have lower life expectancy and higher CVD morbidity. On average, minorities have more limited access to medical care, receive less aggressive care, and receive fewer diagnostic and therapeutic cardiac procedures than non-minority populations. Additionally, most minority groups adhere poorly to prescribed medical regimens and often present to emergency departments rather than primary care physicians for complications of advanced chronic CVD conditions. Thus, research to reduce health disparities by improving CVD outcomes in minorities offers potential for a substantial positive impact on public health. Academic medical centers and institutions that are capable of carrying out such research, however, often lack access to minority patients and have difficulty gaining the trust of those they are able to treat. Minority communities often report greater satisfaction when receiving care from minority providers and are reluctant to receive treatment outside their minority healthcare serving systems.

In general, minorities have high rates of elevated cholesterol, hypertension, cigarette smoking, obesity, metabolic syndrome, and diabetes. Other behavioral, environmental, and occupational risk factors for cardiovascular diseases, such as sleep problems are also common among minorties. These risk factors all contribute to excess CVD morbidity and mortality. Heart failure (HF) is also a major public health problem. The impact of HF on minority populations, such as Native Hawaiians and other Pacific peoples, is unknown. Native Hawaiians are known to have high rates of risk factors for HF and one of the highest rates of CVD mortality in the U.S. The causes of minority health disparities are complex and are not understood completely. Although evidence of genetic, biologic, and environmental factors is well documented, poor outcomes are also attributed to incomplete treatment. Such treatment may be due to limited access to health care or, in some cases, break-down of the medical system or failure of the physician and/or patient to allow for optimal health care, even when access is not impaired. The complex interactions of behavior, socio-economic status (SES), culture, and ethnicity are important predictors of health outcomes and sources of health disparities. Despite efforts to elucidate genetic and environmental risk factors and to promote cardiovascular health in high-risk populations, trends in CVD outcomes suggest that CVD health disparities continue to widen.

The Partnerships Program to Reduce Cardiovascular Health Disparities involves collaboration between research-intensive medical centers (RIMCs) that have a track record of NIH-supported research and patient care and minority healthcare serving systems (MSSs) that lack a strong research program. Each Partnership Program will design and carry out multiple interdisciplinary research projects that investigate complex biologic, behavioral, and societal factors that contribute to CVD health disparities and facilitate clinical research within the MSS. The aim will be to improve CVD outcomes and reduce health disparities. Additionally, each program will provide reciprocal educational and skills development programs to train investigators to conduct research that is aimed at reducing cardiovascular disparities, thereby enhancing research opportunities and enriching cultural sensitivity and cardiovascular research capabilities at both institutions.

The Request for Applications for Partnership Programs to Reduce Cardiovascular Disparities was released in September, 2003. The awards were made in September, 2004.

DESIGN NARRATIVE:

To address heart failure disparities among native Hawaiians and Pacific peoples, a partnership program, the HF Disparities Program (HFD), will be established between the Queen Emma Clinic (QEC) and the Department of Native Hawaiian Health. Partners of the HFD Program include tha following: MedStar Research Institute, Oahu-based Community Health Centers (CHCs), and the Hawaii EXPORT Center, an NIH-funded initiative addressing diabetes-associated disparities in native Hawaiians and Pacific peoples. The HFD Program will address the following aims: determine the reliability and validity of echocardiograms performed by community-based health workers compared to a professionally trained sonographer as the "gold standard"; determine if a culturally competent educational program for heart failure reduces HF hospitalizations and mortality compared to usual care; characterize ethnic differences in the HF syndrome in hospitalized native Hawaiians and Pacific peoples compared to Caucasians; construct HF pedigrees using probands identified at the Queen Emma Clinic for a future HF linkage study in native Hawaiians and Pacific peoples; educate community-based health workers to perform echocardiography scans for the detection of HF in a high risk population of native Hawaiians and Pacific peoples; and train new investigators to conduct research focused on CVD disparities in general, and HF in particular. By achieving these aims, the HFD Program will improve access to HF care at Community Health Centers that serve native Hawaiians and Pacific peoples, fill a gap in knowledge of CVD disparities in native Hawaiians and Pacific peoples, and provide a foundation for future studies on genetic determinants of HF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms and signs of heart failure AND

  1. Left ventricular systolic ejection fraction of less than 40% OR
  2. Left ventricular systolic ejection fraction of less than 60% AND evidence of abnormal diastolic function confirmed by echocardiogram and documented in the patient's medical record
* Discharged from a hospital admission for heart failure as a primary or secondary discharge diagnosis within 6 weeks of study entry
* Self-identified ethnicity/race as Native Hawaiian or Pacific Islander (e.g., Samoan, Tongan, Tahitian, Maori, Marshallese, etc.)

Exclusion criteria

* Heart failure caused by high-output states (i.e., sepsis, etc.) or transient non-cardiac disease
* Terminal illnesses in addition to heart failure (e.g., cancer with projected survival of less than 6 months)
* Currently living in a nursing home
* Currently undergoing hemodialysis or peritoneal dialysis

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be a Native Hawaiian or Pacific Islander (e.g., Samoan, Tongan, Tahitian, Maori, Marshallese, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2004-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Mau, Principal Investigator — University of Hawaii at Manoa; Todd Seto, Principal Investigator — Queen's Medical Center
Locations (2):
- United States (2):
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii at Manoa, Honolulu, Hawaii